CLINICAL TRIAL: NCT01015508
Title: The Role of the Genetic Background Involved in Weight Regain Through Mechanisms Including Energy Expenditure, Physical Activity and Adipogenic Capacity
Brief Title: Adipogenic Capacity as a Mediator of Weight Gain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HumBio_Westerterp09
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
Keywords: Weight loss and maintenance; body composition; energy expenditure; adipogenic capacity; physical activity
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Body Weight Maintenance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High predisposition (Other): High predisposition for weight regain
  Interventions: Other: Very Low Energy Diet (VLED); Other: Weight maintenance
- low predisposition (Other): low predisposition for weight regain
  Interventions: Other: Very Low Energy Diet (VLED); Other: Weight maintenance
- Medium predisposition (Other): Medium predisposition for weight regain
  Interventions: Other: Very Low Energy Diet (VLED); Other: Weight maintenance

INTERVENTIONS:
Other: Very Low Energy Diet (VLED) — a VLED (Modifast) for 2 months in order to reduce body weight
  Other Names: Modifast
Other: Weight maintenance — 10 months

SUMMARY:
To demonstrate differences in response of subjects with a high, low or medium predisposition for weight regain after weight reduction in terms of: body composition; energy expenditure; physical activity; and adipogenic capacity.

DETAILED DESCRIPTION:
The risk for weight regain after weight loss is a major problem for the current obesity treatments, and is largely genetically determined. It is believed that an elucidation of the genetic component in the prognosis of weight management could assist in the development of more effective and individually tailored treatments. However, current research on the genetic component of weight management, and in particular weight regain, is still limited and data available are sometimes inconsistent. The current research proposal aims to identify groups with a high, low or medium predisposition for weight regain, based on a genetic profile and to demonstrate differences in the response of these subjects to a weight maintenance period after weight reduction in terms of body composition, physical activity, adipogenic capacity and energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* BMI 28-35
* healthy, no medication
* no smoking
* stable weight (no weight loss/gain > 5kg in 3 months prior to study)

Exclusion Criteria:

* 28< BMI >35
* use of medication
* smoking
* weight loss/gain > 5kg in 3 months prior to study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | 0, 2 and 12 months

SECONDARY OUTCOMES:
Adipogenic capacity, Physical activity and body composition | 0, 2 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Klaas R Westerterp, Prof, Principal Investigator — Maastricht University
Locations (1):
- Dept. of Human Biology (Maastricht University), Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Camps SG, Verhoef SP, Roumans N, Bouwman FG, Mariman EC, Westerterp KR. Weight loss-induced changes in adipose tissue proteins associated with fatty acid and glucose metabolism correlate with adaptations in energy expenditure. Nutr Metab (Lond). 2015 Oct 24;12:37. doi: 10.1186/s12986-015-0034-1. eCollection 2015. PMID 26500687
- [Derived] Camps SG, Verhoef SP, Westerterp KR. Weight loss-induced reduction in physical activity recovers during weight maintenance. Am J Clin Nutr. 2013 Oct;98(4):917-23. doi: 10.3945/ajcn.113.062935. Epub 2013 Aug 28. PMID 23985804
- [Derived] Verhoef SP, Camps SG, Gonnissen HK, Westerterp KR, Westerterp-Plantenga MS. Concomitant changes in sleep duration and body weight and body composition during weight loss and 3-mo weight maintenance. Am J Clin Nutr. 2013 Jul;98(1):25-31. doi: 10.3945/ajcn.112.054650. Epub 2013 May 22. PMID 23697706
- [Derived] Camps SG, Verhoef SP, Westerterp KR. Weight loss, weight maintenance, and adaptive thermogenesis. Am J Clin Nutr. 2013 May;97(5):990-4. doi: 10.3945/ajcn.112.050310. Epub 2013 Mar 27. PMID 23535105
- [Derived] Verhoef SP, Camps SG, Bouwman FG, Mariman EC, Westerterp KR. Physiological response of adipocytes to weight loss and maintenance. PLoS One. 2013;8(3):e58011. doi: 10.1371/journal.pone.0058011. Epub 2013 Mar 7. PMID 23505452